CLINICAL TRIAL: NCT06452992
Title: Microbiome and Metabolomics Profiling in Children With Obstructive Sleep Apnoea
Brief Title: Microbiome and Metabolomics Profiling in Children With OSA
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kate Ching Ching Chan, Associate Professor, Chinese University of Hong Kong
Other Study IDs: MOSAMM
Record Dates: First submitted 2023-11-01; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine and stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Children aged 6-11 years old with habitual snoring (≥3 nights per week) and PSG confirmed OSA (OAHI of ≥1/hour)
- Controls: Age, sex and BMI matched non-OSA control with PSG confirmed absence of OSA (OAHI < 1 event/h)

SUMMARY:
Objectives: Obstructive sleep apnoea (OSA) exhibits variable susceptibility to end-organ morbidities. Previous studies suggest that physiological sequelae in individuals with OSA promote changes in microbiome, which also interact with metabolic and inflammatory mediators. Therefore, microbiome and metabolomic profiling could potentially reveal the pathological processes underlying OSA. The primary objectives of our study are 1)To investigate the differences in the composition of nasal and stool microbiome between children with OSA and non-OSA controls; 2)To investigate the differences in the urine metabolomic profiles between children with OSA and non-OSA controls.

Hypothesis to be tested: The microbiome composition and urine metabolomic profiles are different between children with OSA and non-OSA controls. Changes in microbiome composition are associated with specific urine metabolomic and inflammatory profiles in children with OSA.

Design and subjects: A prospective case-control study. Chinese children aged 6-11 years old with habitual snoring and polysomnography (PSG) confirmed OSA will be recruited as cases. Non-OSA healthy children will be recruited as controls. All subjects will undergo evaluation including questionnaires, anthropometric measurements, PSG, blood, urine, nasal and stool sampling.

Primary outcome measures: Microbiome and metabolomic profiles in children with OSA compared to non-OSA controls.

Analysis: Comparisons of the microbiome and metabolomic profiles between OSA children and controls. Correlations of microbiome and metabolomic profiles with inflammatory biomarkers and PSG measurements will be evaluated by regression analysis.

Expected results: This study will provide novel data regarding microbiome and metabolomic profiles, and their relationship with inflammatory biomarkers in children with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-11 years old

Exclusion Criteria:

* Previous upper airway surgery, genetic or syndromal disease, congenital or acquired neuromuscular disease, suspected or confirmed congenital or acquired immunodeficiency, known metabolic syndrome, craniofacial abnormalities, structural or congenital heart disease, use of medications or therapy that could affect immunity such as systemic corticosteroids, chemotherapy, radiation therapy, intravenous immunoglobulins.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who attend the Paediatric Respiratory and Sleep Clinic at the Prince of Wales Hospital (PWH) for suspected OSA
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Stool microbiome profiles | 2 years
  Stool microbiome profiles in children with OSA compared to non-OSA controls: MetaPhlAn3 profiles and functional profiling by Functional profiling by HUMAnN3
Urine metabolomic profiles | 2 years
  Urine metabolomic profiles in children with OSA compared to non-OSA controls: hydrophilic and ionic metabolites, lipophilic metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Kate Ching Ching Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided